CLINICAL TRIAL: NCT07154290
Title: A Phase 2 Study to Investigate Ubamatamab With and Without REGN7075 in Treatment-Experienced Participants With Advanced/Metastatic Non-Small Cell Lung Cancer (NSCLC)
Brief Title: A Study to Investigate Ubamatamab With and Without REGN7075 in Adult Participants With Advanced/Metastatic Non-Small Cell Lung Cancer (NSCLC)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R4018-ONC-2476
Record Dates: First submitted 2025-08-26; First posted 2025-09-04 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Advanced/Metastatic Non-Small Cell Lung Cancer
Keywords: NSCLC; Mucin-16 (MUC16); Ubamatamab; Epidermal Growth Factor Receptor (EGFR); REGN7075; Stage IIIB, IIIC or IV
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — sarilumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Arm 1A (Experimental)
  Interventions: Drug: Ubamatamab; Drug: Sarilumab
- Arm 1B (Experimental)
  Interventions: Drug: Ubamatamab; Drug: REGN7075; Drug: Sarilumab
- Arm 1C (Experimental)
  Interventions: Drug: Ubamatamab; Drug: REGN7075; Drug: Sarilumab
- Arm 2A (Experimental)
  Interventions: Drug: Ubamatamab; Drug: Sarilumab
- Arm 2B (Experimental)
  Interventions: Drug: Ubamatamab; Drug: REGN7075; Drug: Sarilumab
- Arm 2C (Experimental)
  Interventions: Drug: Ubamatamab; Drug: REGN7075; Drug: Sarilumab

INTERVENTIONS:
Drug: Ubamatamab — Administered per the protocol
  Other Names: REGN4018
Drug: REGN7075 — Administered per the protocol
  Arms: Arm 1B; Arm 1C; Arm 2B; Arm 2C
Drug: Sarilumab — Administered per the protocol
  Other Names: REGN88SAR153191

SUMMARY:
This study will evaluate two study drugs called ubamatamab and REGN7075, to see if they can help treat advanced or metastatic Non-Small Cell Lung Cancer (NSCLC), and sarilumab, to evaluate to see if it can help with immune-related side effects from ubamatamab.

The study is looking at:

* How well ubamatamab and REGN7075 works
* The side effects that ubamatamab and REGN7075 might cause
* How much ubamatamab and REGN7075 is in the blood at different times
* If the body makes antibodies to ubamatamab and/or REGN7075, this may cause the ubamatamab to not work as well

ELIGIBILITY:
Key Inclusion Criteria:

1. Has histologically or cytologically confirmed diagnosis of advanced (stage IIIB not amenable to definitive chemoradiotherapy or stage IIIC) or metastatic (stage IV) NSCLC
2. Has received appropriate first line standard of care treatment for advanced or metastatic NSCLC, as described in the protocol
3. If platinum doublet chemotherapy was not administered as first line therapy, it is required in a later line of therapy prior to enrollment unless there is a documented reason why it is not appropriate
4. Has tumor tissue (archival or fresh) available for testing MUC16 expression by immunohistochemistry inclusion (IHC), as described in the protocol
5. Has at least 1 radiographically measurable lesion by Computed Tomography (CT) or Magnetic Resonance Imaging (MRI) per RECIST v1.1 criteria. Target lesions may be located in a previously irradiated field if there is documented (radiographic) disease progression in that site
6. Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1

Key Exclusion Criteria:

1. Has progression of disease fewer than 84 days from starting initial anti-Programmed Cell Death (PD)-(L) 1 therapy
2. Experienced toxicity related to prior treatment that has not resolved to grade 1 prior to initiation of study intervention (except alopecia, hearing loss, grade 2 neuropathy, or endocrinopathy managed with hormone replacement therapy)
3. Has untreated or active primary brain tumor, Central Nervous System (CNS) metastases, leptomeningeal disease, or spinal cord compression, as described in the protocol
4. Current participation OR past participation in another investigational study in which an investigational intervention (eg, drug, vaccine, invasive device) was administered within 4 weeks before planned first dose of study intervention in this clinical study
5. Has received prior monoclonal antibody against PD-(L)1 within 21 days of the first dose of study intervention
6. Has had other prior anti-cancer immunotherapy within 21 days prior to study intervention, as described in the protocol
7. Has received prior cytotoxic chemotherapy within 21 days of the first dose of study intervention
8. Has received an anti-EGFR antibody therapy within the following drug-specific window prior to first dose of study intervention (approximately 5 half-lives), as described in the protocol

NOTE: Other protocol defined inclusion / exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-03-18 (Estimated); Primary Completion 2030-06-10 (Estimated); Study Completion 2030-06-10 (Estimated)

PRIMARY OUTCOMES:
Objective response as assessed by the investigator per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 | Up to 5 years

SECONDARY OUTCOMES:
Occurrence of Treatment Emergent Adverse Events (TEAEs) | Up to 5 years
Severity of TEAEs | Up to 5 years
Occurrence of Treatment-Related Adverse Events (TRAEs) | Up to 5 years
Severity of TRAEs | Up to 5 years
Occurrence of Adverse Events of Special Interest (AESIs) | Up to 5 years
Severity of AESIs | Up to 5 years
Occurrence of Serious Adverse Events (SAEs) | Up to 5 years
Severity of SAEs | Up to 5 years
Occurrence of grade ≥2 Cytokine Release Syndrome (CRS) by Lee Criteria | Up to 5 years
Duration of Response (DOR) as assessed by the investigator per RECIST v1.1 | Up to 5 years
Progression-Free Survival (PFS) as assessed by the investigator per RECIST v1.1 | Up to 5 years
Best Overall Response (BOR) of confirmed Complete Response (CR) per RECIST v1.1 | Up to 5 years
Disease Control Rate (DCR) as assessed by the investigator per RECIST v1.1 | Up to 5 years
Incidence of Anti-Drug Antibodies (ADA) to ubamatamab | Up to 5 years
Incidence of ADA to REGN7075 | Up to 5 years
Magnitude of ADA to ubamatamab | Up to 5 years
Magnitude of ADA to REGN7075 | Up to 5 years
Concentrations of ubamatamab in serum | Up to 5 years
Concentrations of REGN7075 in serum | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/